CLINICAL TRIAL: NCT05289960
Title: Lung Ultrasound Score for Prediction of Weaning Outcome
Brief Title: Lung Ultrasound Score and Weaning Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MS-490-2020
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Lung Ultrasound Score; Acute Respiratory Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients eligible for weaning by spontaneous breathing trial (Other)
  Interventions: Other: lung ultrasound
- non invasive ventilation after weaning (Other)
  Interventions: Other: lung ultrasound

INTERVENTIONS:
Other: lung ultrasound — Lung ultrasound score was done at the end of SBT using curved array ultrasound probe 2-5 MHz, Siemens X300, Korea

SUMMARY:
Objectives: Failure of extubation of patients on mechanical ventilation is one of the common problems in the ICU.

Aim of work: To evaluate the validity of lung ultrasound score in prediction of weaning outcomes and post-extubation distress.

DETAILED DESCRIPTION:
Methods: A prospective observational study of 50 patients planned for extubation who passed a spontaneous breathing trial, lung ultrasound score and serum level of NT-PRO BNP were done to all patients at end of spontaneous breathing trial, and all patients were followed after extubation and monitored for oxygenation, re-intubation rate, ICU stay, and ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients age > 18 years

2. Patients intubated and mechanically ventilated for more than 48 hours in the intensive care unit and planned for extubation.

Exclusion Criteria:

* 1. Patients < or =18 years 2. Patients with left ventricular failure

  3. Right ventricular failure

  4. Pulmonary hypertension

  5. Aortic valve disease

  6. Hyperthyroidism

  7. Tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Extubation success | 48 hours
  number of participants that do not need for respiratory support neither NIV nor intubation for one week during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: farouk faris, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt